CLINICAL TRIAL: NCT00782496
Title: A New Contour Blood Glucose Monitoring System With High Frequency Testing Patients
Brief Title: Glucose Meter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTD-2008-09
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Level1 Basic Meter Features (Experimental): Adults with type 1 and type 2 diabetes use only basic features (Level 1) to test their blood. The CONTOUR meter has the basic features such as small meter size, easy to use , No Coding™ technology, 5-second test time, small sample size (0.6 µL), automatic control solution marking, 480 reading memory capacity.
  Interventions: Device: Education + new meter
- Level 2 Advanced Meter Features (Experimental): Adults with type 1 and type 2 diabetes additionally access and use more advanced meter features(Level 2)during blood glucose testing. The advanced features include ability to mark blood glucose values as obtained before or after meals or to set an audible reminder to test.
  Interventions: Device: Education + new meter + feature activation

INTERVENTIONS:
Device: Education + new meter — Diabetes education and a new meter with basic features
  Arms: Level1 Basic Meter Features
Device: Education + new meter + feature activation — Diabetes education and a new meter with advanced features
  Arms: Level 2 Advanced Meter Features

SUMMARY:
The purpose of this study is to evaluate if the meal marker and reminder feature of the Contour meter along with education maintains or increases frequency of testing blood sugar after meals and enables behavioral changes that may lead to improvement in glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with type 1 or type 2 diabetes
2. Persons who are on a pump or are taking at least 1 mealtime injection of insulin a day
3. Persons at least 21 years of age
4. Persons willing to complete all study visits and study procedures including:

   * Using the meal-marker + reminder feature regularly (Group 2 subjects only)
   * Using the paper logbook provided (both Groups)
5. Testing their BG at least 3 times a day during the entire study.
6. Persons who are able to speak, read and understand English
7. Persons who are currently performing self-testing of blood glucose at home routinely (at least 3 times per day) for 4 weeks or more

Exclusion Criteria:

1. Persons who have been using a CONTOUR, BREEZE or BREEZE 2 meter regularly during the previous 6 months
2. Persons who test over 6 times/day regularly
3. Persons who wear a BG sensor 2 weeks or more during each month.
4. Persons with home heath aides who assist with their BG testing.
5. Persons with the following impairments which, in the opinion of the investigator, would seriously compromise the integrity of the study:

   * Significant visual impairment
   * Significant hearing impairment
   * Cognitive disorder
   * Significant unstable co-morbidity (with notable change within the past 3 months)
6. Any other condition as per investigator's discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dace Trence, MD, Principal Investigator — University of Washington Medical Center/Diabetes Care Center; Bruce W Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Ronald Tamler, MD, Phd, MBA, Principal Investigator — Icahn School of Medicine at Mount Sinai; Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (4):
- United States (4):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - International Diabetes Center, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University of Washington Medical Center/Diabetes Care Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Level1 Basic Meter Features: Adults with type 1 and type 2 diabetes using basic meter features
- Level 2 Advanced Meter Features: Adults with type 1 and type 2 diabetes using advanced meter features.
Period: Overall Study
Arm/Group | Level1 Basic Meter Features | Level 2 Advanced Meter Features
Started | 106 | 105
Completed | 92 | 90
Not Completed | 14 | 15
Not completed — Lost to Follow-up | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level1 Basic Meter Features | Level 2 Advanced Meter Features | Total
Number analyzed (Participants) | 106 | 105 | 211
Age, Customized [Median (Full Range); unit: years] | 53 [22 to 81] | 56 [23 to 80] | 55 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 60 | 113
  Male | 53 | 45 | 98
Region of Enrollment [Number; unit: participants]
  United States | 106 | 105 | 211

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Weekly Post-Prandial Blood Glucose Tests Performed by Subjects Using Either Basic or Advanced Meter Features
Time Frame: 6 months
Population: For level 1, 14 subjects were lost to follow-up, that is they did not continue through the study's 4 visits, and data was not available. For level 2, 15 subjects were likewise lost to follow-up and data was not available. For units analyzed, 74 and 68 refer to the number of logbooks available.
Measure: Mean (Standard Error); unit: number of post-prandial tests per week
Arm/Group | Level1 Basic Meter Features | Level 2 Advanced Meter Features
Number analyzed (Participants) | 74 | 68
number of post-prandial tests per week | 7.1 (0.72) | 10.2 (0.72)

2. Secondary Outcome: Percent of Level 2 Participants Who Rated Helpfulness of Advanced Meter Features as 1 or 2
Description: Level 2 participants, who used advanced meter features, responded to questionnaires. They rated helpfulness of the meal marker reminder feature on a 5 point scale, 1 being strongly agree and 5 being strongly disagree.
Time Frame: Over six month period
Population: 63 surveys were available for analysis.
Measure: Number; unit: percent of Level 2 participants
Arm/Group | Level 2 Advanced Meter Features
Number analyzed (Participants) | 63
percent of Level 2 participants | 72.4

ADVERSE EVENTS:
Time Frame: 6 months
Description: All serious adverse events were not linked to the study device.
Arm/Group | Level1 Basic Meter Features | Level 2 Advanced Meter Features
Serious Adverse Events (participants affected / at risk) | 12/106 | 6/105
Other Adverse Events (participants affected / at risk) | 0/94 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level1 Basic Meter Features (N=106) | Level 2 Advanced Meter Features (N=105)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Heart attack (Cardiac disorders) | 1 (1) | 0 (0)
Trachial infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adrenal growth (Endocrine disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diverticulosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mastectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotensive (Cardiac disorders) | 2 (3) | 0 (0)
Lower leg edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coronary artery bypass (Cardiac disorders) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphadema of arm (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less